CLINICAL TRIAL: NCT05264844
Title: The Effects of Two Different Catheter Covers on Patient's Comfort, Satisfaction, Pain Level and Nurse's Satisfaction Randomized Controlled Study"
Brief Title: Peripheral Venous Catheter and Masking Tape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rukiye Burucu, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123456
Record Dates: First submitted 2022-01-19; First posted 2022-03-03 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Personal Satisfaction; Pain; Comfort
Keywords: Peripheral venous catheter; chemotherapy; patch; fixation
MeSH Terms: conditions — Personal Satisfaction; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Only the statistician will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- masking tape group (Experimental): Masking tape will be used
  Interventions: Other: Masking tape
- standard catheter dressing group (No Intervention): Medical plaster to be used (It is routine practice in the clinic.)

INTERVENTIONS:
Other: Masking tape — IV catheters will be fixed with masking tape
  Arms: masking tape group

SUMMARY:
urpose: This study will be carried out to determine the effect of two different catheter covers on the comfort, satisfaction, pain level of the patient and the satisfaction of the nurse.

Materials and Methods: This study, which is planned as an open-label randomized controlled post-test study, will be carried out between December 2021 and February 2022. Data; Descriptive Properties will be collected with the Information Form and Visual Analog Scale (Visual Analog Scale-VAS). Data will be collected face to face by researchers.

DETAILED DESCRIPTION:
Peripheral venous catheter (PVK) is applied to patients who apply to the hospital due to outpatient chemotherapy and need to receive treatment by intravenous route. This application is carried out by nurses. During their education, nurses receive theoretical and practical training on PVC applications. Nurses; They are the primary health professionals who are responsible for determining the PVC site, deciding on the catheter number to be used, applying the correct technique, performing the recommended intravenous (IV) interventions, following the complications that may develop by performing the necessary controls, ensuring the continuity of the application and providing catheter care.

The effective application of interventions such as transfusion of intravenous fluids, chemotherapy drugs, blood and blood products, and total parenteral feeding in cancer patients is provided by PVK. The application of PVC is a necessity for the treatment of the individual receiving treatment and may cause pain, deterioration in comfort and dissatisfaction. Although the widespread use of peripheral venous catheters provides great benefits, it has been reported that undesirable events such as phlebitis, infiltration, obstruction, leakage, and rarely infection occur when applied incorrectly and inadequately. In order for peripheral venous catheters to be used effectively in treatment, it is important to fix them with the correct technique. Detection becomes more important in the use of chemotherapy agents. The patches used for fixation adhere to the glove and are difficult to remove from the patient's skin. Therefore, both the nurse and the patient feel discomfort. For this reason, it would be appropriate to use a material that can be easily torn off with a glove, does not adhere to the glove, and fixes the patient's catheter well. This product should also be able to be easily removed without harming the patient's skin.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being open to communication and cooperation
* Being conscious and able to answer questions
* Volunteering for research
* Being receiving chemotherapy treatment with a peripheral venous catheter

Exclusion Criteria:

* Having a disease that may affect the ability to make decisions (dementia, psychological disorders, etc.)
* Having sensory losses such as vision and hearing
* Being in terminal period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Pain level | a week
  To be evaluated with "Visual analog scale"
Patient comfort | a week
  To be evaluated with "Visual analog scale"
Nurse's practice satisfaction | a week
  To be evaluated with "Visual analog scale"

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Univercity, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided